CLINICAL TRIAL: NCT04511624
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled, Single Subcutaneous or Intravenous Ascending Dose Trial to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of IBI112 in Healthy Subjects
Brief Title: Single Dose Tolerability and Pharmacokinetics of IBI112 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI112A101
Record Dates: First submitted 2020-08-03; First posted 2020-08-13 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): IBI112 SC dose1
  Interventions: Drug: IBI112 dose1
- Cohort 2 (Experimental): IBI112 SC dose2
  Interventions: Drug: IBI112 dose2
- Cohort 3 (Experimental): IBI112 SC dose3
  Interventions: Drug: IBI112 dose3
- Cohort 4 (Experimental): IBI112 IV dose4
  Interventions: Drug: IBI112 dose4
- Cohort 5 (Experimental): IBI112 IV dose3
  Interventions: Drug: IBI112 dose5
- Cohort 6 (Experimental): IBI112 SC dose5
  Interventions: Drug: IBI112 dose6
- Cohort 7 (Experimental): IBI112 IV dose5
  Interventions: Drug: IBI112 dose7

INTERVENTIONS:
Drug: IBI112 dose1 — Drug: IBI112 SC dose1 Drug:placebo
  Arms: Cohort 1
Drug: IBI112 dose2 — Drug: IBI112 SC dose2 Drug:placebo
  Arms: Cohort 2
Drug: IBI112 dose3 — Drug: IBI112 SC dose3 Drug:placebo
  Arms: Cohort 3
Drug: IBI112 dose4 — Drug: IBI112 SC dose4 Drug:placebo
  Arms: Cohort 4
Drug: IBI112 dose5 — Drug: IBI112 IV dose5 Drug:placebo
  Arms: Cohort 5
Drug: IBI112 dose6 — Drug: IBI112 SC dose6 Drug:placebo
  Arms: Cohort 6
Drug: IBI112 dose7 — Drug: IBI112 IV dose7 Drug:placebo
  Arms: Cohort 7

SUMMARY:
This is a the first in human study to evaluate the safety, tolerability, PK and PD of single subcutaneous or intravenous dose of IBI112 in healthy subjects

DETAILED DESCRIPTION:
In this first in human, phase 1, randomized, double-blind, placebo-controlled study, a single subcutaneous or intravenous dose of IBI112 will be administered to 46 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female 18 to 45 years of age at the time of consent
2. BMI of 19-26Kg/m2 and weight of 50-100kg
3. Must provide written informed consent, and in the investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements

Exclusion Criteria:

1. Subjects who have a medical history of liver, kidney, cardiovascular, nervous / mental, gastrointestinal, respiratory, urinary, endocrine
2. Subjects who have a history of relapse or chronic infection, or a history of acute infection within 2 weeks;
3. Subjects who have previously used anti-IL-12 / 23 or anti-il-23 drugs;
4. Subjects who have clinically significant abnormalities determined by vital signs, physical examination, and laboratory measurements;
5. Subjects who are not suitable for this trial due to other reasons In the investigator' opinion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events in healthy volunteers with single ascending doses of IBI112 | Day1 to Day 113 post dose

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) - Pharmacokinetic Assessment | Day 113
  IV dose & SC dose
Time to Maximum Concentration (Tmax) - Pharmacokinetic Assessment | Day 113
  SC dose
Area Under the Curve Extrapolated to Infinity (AUC0-∞) - Pharmacokinetic Assessment | Day 113
  IV dose & SC dose
Half-Life (t1/2) - Pharmacokinetic Assessment | Day 113
  IV dose & SC dose
Volume of Distribution (Vd) - Pharmacokinetic Assessment | Day 113
  IV dose & SC dose

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China

REFERENCES:
- [Derived] He J, Du W, Yang H, Wang J, Cai C, Ma Q, Li N, Yu J, Wu X, Wu J, Chen Y, Cao G, Zhang J. Safety and pharmacokinetics of IBI112, an IL-23 monoclonal antibody, in Chinese healthy volunteers: a first-in-human phase 1 study. Expert Opin Investig Drugs. 2023 Jul-Dec;32(7):669-675. doi: 10.1080/13543784.2023.2230122. Epub 2023 Jun 29. PMID 37358916